CLINICAL TRIAL: NCT01612351
Title: Multimodality Risk Adapted Therapy Including Carboplatin/Paclitaxel/Lapatinib as Induction for Squamous Cell Carcinoma of the Head and Neck Amenable to Transoral Surgical Approaches
Brief Title: Multimodality Risk Adapted Tx Including Induction Chemo for SCCHN Amenable to Transoral Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1125
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and neck cancer; Squamous Cell Carcinoma; Phase II; Transoral Surgery; Induction Chemotherapy; Carboplatin; Paclitaxel; Lapatinib
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Carboplatin; Paclitaxel; Lapatinib; Cisplatin; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-Randomized Single-Arm (Experimental): All participants will receive induction chemotherapy and transoral surgery. Following surgery, participants will be stratified into a risk category (low, medium, or high). Subjects in the low risk category will receive no further treatment after their transoral surgery. Subjects in the medium risk category will receive ipsilateral radiation concurrent with weekly cisplatin, and subjects in the high risk category will receive cisplatin every three weeks with concurrent bilateral radiation.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Lapatinib; Drug: Cisplatin; Radiation: Ipsilateral Radiation; Radiation: Bilateral Radiation; Procedure: Transoral Surgery

INTERVENTIONS:
Drug: Carboplatin — Weekly carboplatin given intravenously for 6 weeks during induction chemotherapy.
  Other Names: Paraplatin
Drug: Paclitaxel — Weekly paclitaxel given intravenously prior to carboplatin infusion for 6 weeks during induction chemotherapy.
  Other Names: Taxol
Drug: Lapatinib — Lapatinib (1000mg) taken by mouth once a day either one hour before or one hour after a meal for 6 weeks during induction chemotherapy. Participants deemed high risk following transoral surgery will additionally take lapatinib daily concurrently with their chemoradiation therapy.
  Other Names: Tykerb
Drug: Cisplatin — Weekly cisplatin given intravenously for 6 weeks concurrent with ipsilateral radiation. Alternative regimens may be substituted for cisplatin in patients who are not candidates for cisplatin at the discretion of the investigator. If carboplatin is used, a maximum of 125 mL/min must be used, as per standard of care.
  Other Names: Platinol
Drug: Cisplatin — Cisplatin given once every 3 week cycle intravenously for 5-7 weeks concurrent with bilateral radiation and daily lapatinib. Alternative regimens may be substituted for cisplatin in patients who are not candidates for cisplatin at the discretion of the investigator. If carboplatin is used, a maximum of 125 mL/min must be used, as per standard of care.
  Other Names: Platinol
Radiation: Ipsilateral Radiation — After transoral surgery, subjects deemed medium risk will receive ipsilateral radiation as per standard of care 5 days/week for 6 weeks concurrent with weekly cisplatin.
  Other Names: Radiation therapy
Radiation: Bilateral Radiation — After transoral surgery, subjects deemed high risk will receive bilateral radiation as per standard of care 5 days/week for 5-7 weeks concurrent with cisplatin every 3 weeks and daily lapatinib.
  Other Names: Radiation therapy
Procedure: Transoral Surgery — Transoral resection by robotic or microscopic approach, which will be at the discretion of the treating surgeon.
  Other Names: Surgery

SUMMARY:
The purpose of this study is to see if a three method risk adapted design using induction chemotherapy, transoral surgery and radiation chemotherapy will lessen toxic effects and make treatment of squamous cell carcinoma of the head and neck (SCCHN) better.

DETAILED DESCRIPTION:
This is a single-arm non-randomized two-stage phase II trial in previously untreated patients with squamous cell carcinoma of the head and neck (SCCHN) arising in the oral cavity, oropharynx, or supraglottic larynx amenable to a transoral surgical approach. Treatment will consist of 3 parts: neoadjuvant induction with weekly carboplatin and paclitaxel in combination with daily lapatinib for 6 weeks (PART 1) prior to transoral surgery (PART 2). Post-operative treatment (PART 3) will vary depending on the risk category assigned to the patient following surgery as follows: no further treatment or treatment limited to involved field radiation (low risk), ipsilateral radiation concurrent with weekly chemotherapy ( medium risk); or cisplatin every 3 weeks and daily lapatinib concurrent with bilateral radiation (high risk).

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically proven primary squamous cell carcinoma arising in the oral cavity, oropharynx, or supraglottic larynx, and amenable to transoral approach
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (see Appendix C)
* Measurable disease as per Response Evaluation Criteria In Solid Tumors (RECIST1.1)
* Age ≥18 years
* Adequate bone marrow function as demonstrated by: Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3; Hgb > 10 g/dL (use of transfusion to reach this threshold prior to study initiation is acceptable); Platelet count ≥ 100,000/mm3
* Adequate hepatic and renal function as demonstrated by: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN); Total serum bilirubin ≤1.5 mg/dL; Creatinine clearance (CrCL) ≥ 40ml/min as measured via Cockcroft-Gault
* Left ventricular ejection fraction (LVEF) must be > the lower limit of normal (LLN) per institutional standards by either echocardiography or radionuclide-based multiple gated acquisition (MUGA)
* Negative serum human chorionic gonadotropin (β-hCG) pregnancy test within 72 hours of day 1 of induction chemotherapy in women of child-bearing potential
* All males and females of childbearing potential must agree to use adequate contraception during the study. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Signed an institutional review board (IRB)-approved informed consent document for this protocol.

Exclusion Criteria:

* tumor 1-node 0 (T1N0) disease or tumor 2-node 0 (T2N0) disease
* Any metastatic disease
* Not considered eligible for any of the chemotherapy agents included in the induction regimen.
* Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Major surgery within 3 weeks prior to day 1 of study treatment from which the patient has not completely recovered
* Current use of a prohibited medication or requires any of these medications during treatment with lapatinib prior to study entry
* Receiving any investigational agent currently, or within 2 weeks of Day 1 of treatment on this study
* Active, serious infection, medical, or psychiatric condition that would represent an inappropriate risk to the patient or would likely compromise achievement of the primary study objective, including unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction ≤ 6 months prior to study entry
* Adequate swallowing function or gastric-tube for drug administration. Of note, lapatinib can be administered via G-tube in a slurry for patients who cannot swallow
* Other prior or concomitant malignancies with the exception of: Non-melanoma skin cancer; In-situ malignancy; Low-risk prostate cancer after curative therapy; Other cancer for which the patient has been disease free for ≥ 3 years
* Pregnant or lactating women, or adults of reproductive potential who do not agree to use adequate contraception during study treatment (see definition of adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2025-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Chemotherapy Followed by Transoral Surgery: All participants will receive induction chemotherapy and transoral surgery. Following surgery, participants will be stratified into a risk category (low, medium, or high). Subjects in the low risk category will receive no further treatment after their transoral surgery. Subjects in the medium risk category will receive ipsilateral radiation concurrent with weekly cisplatin, and subjects in the high risk category will receive cisplatin every three weeks with concurrent bilateral radiation.
Period: Chemotherapy
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Started | 40
Completed | 40
Not Completed | 0
Period: Transoral Surgery
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Started | 39 (One patient completed chemotherapy then withdrew before surgery.)
Completed | 39
Not Completed | 0
Period: Post-Operative Treatment
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Started | 39
Completed | 39 (One patient completed chemotherapy then withdrew before surgery.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40
Disease Location [Count of Participants; unit: Participants]
  Supraglottic Larynx | 5
  Oral Cavity | 4
  Hypopharynx | 1
  Oropharynx | 30
Stage of disease [Count of Participants; unit: Participants] — Anatomic stage for NSCLC is the American Joint Committee on Cancer (AJCC) primary tumor, regional nodes, metastasis (TNM) system, which is based on:
  Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Once the categories have been determined, this information is combined into a prognostic group. Higher numbers mean the cancer is more advanced. N1- 1 lymph node on the same side as the original tumor. N2a- Spread to 1 lymph node on the same side. N2b- spread to 2 or more lymph nodes on same side. N2c- 1 or more lymph nodes on both sides.
  Participants
    T1N1 | 1
    T1N2a | 4
    T1N2b | 6
    T2N1 | 4
    T2N2a | 5
    T2N2b | 12
    T2N2c | 2
    T3N0 | 3
    T3N2c | 1
    T4N1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Evaluation of target lesions through tumor imaging (CT scan, MRI, and/or chest x-ray) at 3-5 weeks post induction chemotherapy. Overall response rate will be based on RECIST criteria. Overall response rate (ORR) is defined as the number of patients who have a partial or complete response to therapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 11 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Number analyzed (Participants) | 40
Participants | 37

2. Secondary Outcome: Feasibility of 3 Part Therapy
Description: Percentage of patients successfully completing 3 part therapy will be used to assess the feasibility of 3 part therapy consisting of induction chemotherapy, surgery, and risk-adapted use of chemoradiation.
Time Frame: 2 years
Population: All participants started to receive study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Number analyzed (Participants) | 40
Participants
  completed | 39
  not-completed | 1

3. Secondary Outcome: Number of Patients Who Decreased in Risk Level Post Induction Chemotherapy.
Description: Number of patients who no longer need radiation (have decreases in risk level post induction therapy). Estimations of Risk level pre-induction will be based on physical examination and imaging, post-induction risk level will be determined based on pathologic evaluation or surgical specimen.
Time Frame: 11 weeks
Population: One patient withdrew before surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Number analyzed (Participants) | 39
Participants | 29

4. Secondary Outcome: Overall Survival
Description: Overall survival is measured from the time the patient goes on treatment until death.
Time Frame: 15 years
Reporting Status: Not Posted

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival associated with 3 part therapy consisting of induction chemotherapy, surgery and risk-adapted use of chemoradiation. Defined as per RECIST criteria. Physical examination, imaging of target lesions by CT scan or MRI and chest imaging (CT or Chest x-ray, if clinically indicated) every 3 months (+/- 30 days) for 18 months following end of treatment. "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 15 years
Reporting Status: Not Posted

6. Secondary Outcome: Voice and Swallowing Function- MD Anderson Dysphagia Inventory (MDADI)
Description: The MD Anderson Dysphagia Inventory (MDADI) is a 20 item assessment designed to measure voice and swallowing function. Participants were asked 13 symptom questions and 6 interference items (walking, working) and asked id the 1- strongly agree to 5 strongly disagree. Scores were summed for a range of 20-100. The lower the score the worse the outcomes.
Time Frame: Pre-treatment up to 1 year post surgery
Population: Subjects were encouraged to complete the assessments but it was left to their discretion. Participants with data available reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-treatment; Post-Induction; 1 Year Post Surgery: All participants will receive induction chemotherapy and transoral surgery. Following surgery, participants will be stratified into a risk category (low, medium, or high). Subjects in the low risk category will receive no further treatment after their transoral surgery. Subjects in the medium risk category will receive ipsilateral radiation concurrent with weekly cisplatin, and subjects in the high risk category will receive cisplatin every three weeks with concurrent bilateral radiation.
Arm/Group | Pre-treatment | Post-Induction | 1 Year Post Surgery
Number analyzed (Participants) | 39 | 25 | 26
units on a scale | 83.90 (14.04) | 86.26 (13.24) | 81.90 (16.56)

7. Secondary Outcome: Voice and Swallowing Function - Voice-Related Quality of Life Assessment (VRQOL)
Description: The Voice-Related Quality of Life Tool is a 10 item list of possible voice-related problems. The participant answers 1-5 with 1 being none, not a problem to 5, problem is as bad as it can be. An algorithm is used to calculate the scores, so that sum scores range from 0 to 100, where 0 indicates poor V-RQOL and 100 indicates good V-RQOL
Time Frame: Pre-treatment up to 1 year post surgery
Population: Patients were encouraged to complete the assessment but at their discretion. Participants with data available reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-treatment | Post-Induction | 1 Year Post Surgery
Number analyzed (Participants) | 38 | 25 | 23
units on a scale | 93.42 (13.20) | 92.00 (20.12) | 91.85 (13.80)

8. Secondary Outcome: Estimate the Pathologic Complete Response Rate at the Primary Site and in the Neck Following Induction Chemotherapy
Description: Pathologic complete response (pCR) is the disappearance of all signs of cancer in tissue samples removed during surgery or biopsy (pT0). Also called pathologic complete remission. Pathologic Partial Response (pPR), is the presence of only non-invasive cancer in tissue samples (<pT2)
Time Frame: 11 weeks
Population: All participants received induction chemotherapy and underwent surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Number analyzed (Participants) | 39
Participants
  Pathologic complete response (pCR) | 14
  Pathologic Partial Response (pPR) | 25

9. Secondary Outcome: Response Rates at the Primary Site
Description: Evaluation of target lesions through tumor imaging (CT scan, MRI, and/or chest x-ray) at 3-5 weeks post induction chemotherapy. Overall response rate will be based on RECIST criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 11 weeks
Population: All participants received induction chemotherapy and radiological tumor response evaluation was completed.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Randomized Single-Arm: All participants will receive induction chemotherapy and response evaluation was completed.
Arm/Group | Non-Randomized Single-Arm
Number analyzed (Participants) | 39
Participants
  Complete Response | 15
  Partial Response | 21
  Stable Disease | 3

10. Secondary Outcome: Number of Subjects Who Experience Grade 3/4 Adverse Events According to CTCAE 4.0
Description: The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Number analyzed (Participants) | 40
Participants
  Alanine aminotransferase increased | 2
  Aspartate Aminotransferase increased | 1
  Chest pain- cardiac | 1
  Diarrhea | 5
  Fatigue | 4
  Febrile neutropenia | 4
  Hyperglycemia | 1
  Hyponatremia | 1
  Hypotension | 1
  Lymphocyte count decreased | 1
  Nausea | 1
  Neutrophil count decreased | 22
  Palmar-plantar erythrodysesthesia syndrome | 1
  Peripheral sensory neuropathy | 2
  Rash acneiform | 4
  Sepsis | 1
  White blood cell decreased | 15

11. Secondary Outcome: the Kinome Response to Induction Chemotherapy
Description: Describe the kinome response to induction chemotherapy (lapatinib, paclitaxel, and carboplatin) in patients who consent to this optional evaluation via co-enrollment in LCCC0121
Time Frame: 11 weeks
Population: The data were unable to be analyzed because co-enrollment with LCCC0121 could not be implemented.
Groups:
- Induction Chemotherapy Followed by Transoral Surgery: All participants received LCCC1125 study treatment and co-enrolled with o-enrollment with the LCCC0121 study.
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
Number analyzed (Participants) | 0

12. Secondary Outcome: Response Rates at the Neck.
Description: Evaluation of target lesions through tumor imaging (CT scan, MRI, and/or chest x-ray) at 3-5 weeks post induction chemotherapy. Overall response rate will be based on RECIST criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for neck lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 11 weeks
Population: All participants received induction chemotherapy and radiological tumor response evaluation was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Randomized Single-Arm
Number analyzed (Participants) | 29
Participants
  Complete Response | 11
  Partial Response | 15
  Stable Disease | 3

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Induction Chemotherapy Followed by Transoral Surgery
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Chemotherapy Followed by Transoral Surgery (N=40)
Chest pain - cardiac (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Chemotherapy Followed by Transoral Surgery (N=40)
Abdominal pain (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 12
Anemia (Blood and lymphatic system disorders) | 25
Anorexia (Metabolism and nutrition disorders) | 5
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Aspartate aminotransferase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 6
Blurred vision (Eye disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 12
Creatinine increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 5
Diarrhea (Gastrointestinal disorders) | 28
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 10
Dyspepsia (General disorders) | 3
Edema face (General disorders) | 2
Edema limbs (General disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 20
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypotension (Vascular disorders) | 3
Insomnia (Psychiatric disorders) | 4
Lymphocyte count decreased (Investigations) | 10
Mucositis oral (Gastrointestinal disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Nausea (Gastrointestinal disorders) | 22
Neutrophil count decreased (Investigations) | 31
Oral pain (Gastrointestinal disorders) | 2
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 14
Platelet count decreased (Investigations) | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 18
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
White blood cell decreased (Investigations) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes